CLINICAL TRIAL: NCT03977441
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study: Evaluation of the Efficacy and Safety of Agomelatine in the Treatment of Sleep Disorders and Depression in Patients With Parkinson's Disease
Brief Title: the Efficacy and Safety of Agomelatine in the Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chun-Feng Liu, Professor, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JD-LK-2019-008-02
Record Dates: First submitted 2019-05-12; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Parkinson Disease; Depression; Sleep Disorders; Circadian Rhythm Disorders
MeSH Terms: conditions — Parkinson Disease; Depression; Sleep Wake Disorders; Chronobiology Disorders | interventions — agomelatine; Pramipexole

STUDY DESIGN:
Intervention Model Description: treatment group: treated with agomelatine control group: treated with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind placebo control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): treated with Pramipexole 0.75mg/d（0.25mg tid)+placebo 25mg qn *2weeks than Pramipexole 0.75mg/d（0.25mg tid)+placebo 50mg qn * 10 weeks
  Interventions: Drug: Agomelatine or PIacebo
- experimental group (Experimental): treated with Pramipexole 0.75mg/d（0.25mg tid)+Agomelatine25 mg qn *2weeks than Pramipexole 0.75mg/d（0.25mg tid)+Agomelatine 50mg qn * 10weeks
  Interventions: Drug: Agomelatine or PIacebo

INTERVENTIONS:
Drug: Agomelatine or PIacebo — control group:Pramipexole+pIacebo experimental group:Pramipexole+Agomelatine
  Other Names: Pramipexole

SUMMARY:
Among the patients with Parkinson's disease, about 40%~50% will suffer from depression, 40% will suffer from anxiety, and 40%~60% will suffer from sleep disorder. These non-motor symptoms of Parkinson's disease will cause great physical and psychological pain and affect the quality of life seriously. Commonly used therapeutic drugs, such as selective serotonin reuptake inhibitor (SSRI) and clonazepam, can cause a variety of side effects, including serotonin syndrome, sexual dysfunction, daytime fatigue, insomnia, residual effects and increased risk of falls. Therefore, a new and more reasonable therapeutic choice should be sought. Agomelatine is a new type of antidepressant with novel mechanism, and can improve sleep structure and circadian rhythm. The aim of this multi-center randomized controlled trial (RCT) is to clarify the role of agomelatine in improving sleep disorders and depression in patients with Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as Parkinson's disease conforming to 2015 International Movement Disorder Society(MDS) diagnostic criteria
* Hoehn-Yahr ≤ 3 at "open" stage
* Mini-mental State Examination(MMSE) ≥ 24 points;
* Pittsburgh Sleep Quality Index (PSQI) > 7 points;
* HAMD-17 > 13 points
* Pramipexole hydrochloride tablets 0.75mg / d (0.25mg tid) has been used stably for one month
* Signed informed consent

Exclusion Criteria:

* Parkinson's syndrome and Parkinsonism-Plus syndrome
* Parkinson's movement symptoms are still fluctuating or the treatment of Parkinson's movement symptoms is unstable
* Hepatitis B virus carriers/patients, hepatitis C virus carriers/patients, patients with impaired liver function or elevated transaminase levels above the upper limit
* Other serious neurological diseases, mental illnesses and physical illnesses
* History of alcohol and drugs dependence
* Dementia
* Combined treatment with CYP1A2 strong inhibitor (fluvoxamine, ciprofloxacin, rifampicin, amiodarone, mexiletine, atazanavir, etc.)
* High suicide risk or suicide attempt within 6 months (third item of HAMD-17 ≥ 3)
* Antidepressant medication or other psychiatric treatment in the past month
* pregnant or lactating
* intolerance or allergy to agomelatine active ingredients and excipients
* other conditions that are not suitable for the study considered by the investigators

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of the treatment on the sleep disorders in Parkinson's disease evaluated by PSQI scale score change | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  The Pittsburgh sleep quality index (PSQI) is a widely used sleep evaluation scale in the Chinese population. The sensitivity and specificity of the PSQI (cut-off at 7) are 98.3% and 90.2%, respectively. PSQI has been used to evaluate the sleep disorders in patients with Parkinson's disease focusing on their sleep habits primarily.

SECONDARY OUTCOMES:
The efficacy of the treatment on the sleep disorders in Parkinson's disease evaluated by PDSS, sleep diary and activity trackers | PDSS:visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week); Sleep diary and activity trackers: 12 weeks, through study completion.
  The Parkinson disease sleep scale (PDSS) is used to analyze the underlying causes of sleep disorders based on the results of each factor. In 2010, the International Movement Disorder Society (MDS) recommended that both PDSS and PSQI can be used for the screening and assessment of sleep disorders in the Parkinson's disease.
  Sleep diary is an internationally recognized method to assist the examination of sleep disorders, and keeping recording a sleep diary every day is an effective therapy for some patients with insomnia.
  Activity trackers can monitor and track fitness-related metrics such as distance walked or run, calorie consumption, heartbeat and quality of sleep, which can be used as a reference of patients' sleep quality and circadian rhythm.
The efficacy on the excessive daytime sleepiness of patients with Parkinson's disease | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  Scale: Epworth sleepiness scale(ESS) score change The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'. The questionnaire takes no more than 2 or 3 minutes to answer.
The efficacy on the fatigue of patients with Parkinson's disease | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  Scale:The Fatigue Severity Scale (FSS) score change The Fatigue Severity Scale (FSS) is a scale used in the evaluation of fatigue that affects patients. A list of statements/questions is provided. These statements are related to the different aspects of fatigue and how it affects the body. While rating the questions, one should make use of the scale with numbers from 1 to 7. If a person strongly agrees with a particular statement, the rating of 7 should be given. Strong disagreement is expressed by rating the question as 1. The sum total of ratings given to all questions is used to determine the degree or severity of fatigue that a person is suffering from. The total score of 36 or above calculated using the scale indicates that a person is suffering from fatigue-related health problem. A score that is lower than 36 shows that the health is normal.
The efficacy on the circadian rhythm of patients with Parkinson's disease | visit1(baseline),visit3(6th week),visit4(12th week)
  Scale: The Morningness-Eveningness Questionnaire (MEQ) score change Circadian rhythm disorder is a kind of important sleep disorder. Body temperature and hormone level changes are effective methods to determine the daily cycle, but these methods are cumbersome. The scale evaluation is much easier to implement. The Morningness-Eveningness Questionnaire (MEQ) is the most widely known questionnaire to assess circadian preference. Cut-off points were evaluated: a range of 14-52 for Evening types, 53-64 for neither types, and 65-86 for Morning types.
The efficacy on the rapid eye movement sleep behavior disorder (RBD) of patients with Parkinson's disease | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  Scale: The Rapid Eye Movement Sleep Behavior Disorder Questionnaire-Hong Kong (RBDQ-HK) score change It has been reported that the incidence of RBD in nucleoproteins disease is 90% for multiple system atrophy (MSA) and 38-56% for Parkinson's disease (PD). Therefore, the proportion and severity of RBD in the Parkinson's disease were needed to screened through the RBD screening questionnaire. The rapid eye movement sleep behavior disorder questionnaire (RBDQ)-Hong Kong was the first tool developed for quantifying the severity of RBD. The RBDQ-HK is a self-administered questionnaire with 13 questions. The RBDQ-HK score can range from 0 to 100. The sum total of ratings given to all questions is used to determine the degree or severity of RBD that a person is suffering from. The higher the RBDQ-HK score is, the worse the symptoms are.The best cut-off score was 17/18.
The efficacy on the depression of patients with Parkinson's disease | visit1(baseline),visit3(6th week),visit4(12th week)
  Scales: The Hamilton Depression Scale-17 (HAMD-17) score change The Hamilton Depression Scale (HAMD) is a test measuring the severity of depressive symptoms in individuals, often those who have already been diagnosed as having a depressive disorder.In the 17-item version, nine of the items are scored on a five-point scale, ranging from 0 (not present) to 4 (severe). The remaining eight items are scored on a three-point scale, from 0 to 2, with zero representing absence of symptom, one indicating doubt that the symptom is present, and two representing clear presence of symptoms. Scores can range from 0 to 54. One formulation suggests that scores between 0 and 6 indicate a normal person with regard to depression, scores between 7 and 17 indicate mild depression, scores between 18 and 24 indicate moderate depression, and scores over 24 indicate severe depression.
The efficacy on the anxiety of patients with Parkinson's disease | visit1(baseline),visit3(6th week),visit4(12th week)
  Scales: The Hamilton Anxiety Scale(HAMA) score change
  The Hamilton Anxiety Scale(HAMA) is a widely used interview scale to measure the severity of a patient's anxiety, based on 14 parameters, including anxious mood, tension, fears, insomnia, somatic complaints and behavior at the interview. The major value of HAM-A is to document the results of pharmaco- or psychotherapy, rather than as a diagnostic or screening tool. It takes 15-20 minutes to complete the interview and scoring. Each item is simply given a 5-point score: 0 (not present) to 4 (severe). The HAMA score can range from 0 to 56. The best cut-off score was 14.
The efficacy on the movement of patients with Parkinson's disease | visit1(baseline),visit3(6th week),visit4(12th week)
  Scale: Unified Parkinson's Disease Rating Scale (UPDRS-III) score change The European Medicines Agency (EMA) guideline mentions the UPDRS II and III scales as accepted scales to measure the efficacy of a drug for Parkinson's Disease. The Unified Parkinson's Disease Rating Scale-III (UPDRS-III) is the most widely used scale currently available for the clinical evaluation of motor dysfunction in Parkinson's disease (PD). Each item is simply given a 5-point score: 0 (Absent) to 4 (Marked in amplitude and present most of the time). The UPDRS-III score can range from 0 to 56. The higher the UPDRS-III score is, the worse the symptoms are.
The efficacy on the life quality of patients with Parkinson's disease | visit1(baseline),visit3(6th week),visit4(12th week)
  Scale: Parkinson's Disease Questionnaire-8 (PDQ-8) score change Substantial evidence is available to suggest that the Parkinson's Disease Questionnaire (PDQ) is reliable, valid, responsive, acceptable and feasible as the tool for the assessment of quality of life in Parkinson's disease patients. For these reasons it has been widely adopted and generally considered the industry 'gold standard'. The PDQ is available in the 39-point PDQ-39 or the short form PDQ-8 (8 items). The PDQ-8 contains eight of the original 39 items of the PDQ-39; one item selected from each of the 8 scales.The PDQ-8 provides a reliable measure of overall health status and is ideal for studies in which a shorter questionnaire is preferred. Each item is simply given a 5-point score: 0 (Absent) to 4 (present most of the time). The PDQ-8 score can range from 0 to 32. The higher the PDQ-8 score is, the worse the symptoms are.
Dosage and frequency of sedative and hypnotic drugs | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  Record the dosage and frequency of sedative and hypnotic drugs taken by the patients every visit and analyze the difference between two groups
The Safety of Agomelatine in the Patients With Parkinson's Disease - the effect on the total number of red blood cells. | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  The total number of red blood cells will be monitored through the blood routine examination to see whether the number will change abnormally.
  Normal range of the total number of red blood cells is 4.0-5.50*10^12/L (male) and 3.5～5.0*10^12/L (female) (reference value range)
The Safety of Agomelatine in the Patients With Parkinson's Disease - the effect on the total number of white blood cells. | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  The total number of white blood cells will be monitored through the blood routine examination to see whether the number will change abnormally.
  Normal range of the total number of white blood cells is 4-10*10^9/L (male) and 4-10*10^9/L (female) (reference value range)
The Safety of Agomelatine in the Patients With Parkinson's Disease - the effect on the platelet count. | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  The platelet count will be monitored through the blood routine examination to see whether the number will change abnormally.
  Normal range of the platelet count is 100-300*10^9/L (male) and 100-300*10^9/L (female) (reference value range)
The Safety of Agomelatine in the Patients With Parkinson's Disease - the effect on the concentration of the hemoglobin. | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  The concentration of the hemoglobin will be monitored through the blood routine examination to see whether it will change abnormally.
  Normal range of the concentration of the hemoglobin is 120-160*g/L (male) and 110-150*g/L (female) (reference value range)
The Safety of Agomelatine in the Patients With Parkinson's Disease - the effect on the liver function | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  the liver function will be monitored through the examination of the alanine aminotransferase (ALT) and the aspartate aminotransferase (AST) in the biochemical routine examination Normal range of the concentration of the ALT is 0～40U/L (reference value range) Normal range of the concentration of the AST is 0～40U/L (reference value range)
The Safety of Agomelatine in the Patients With Parkinson's Disease - the effect on the renal function | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  the renal function will be monitored through the examination of the creatinine (Cr) and the urea nitrogen (BUN) in the biochemical routine examination Normal range of the concentration of the Cr is 53～106umol/L (male) and 44～97umol/L (female) (reference value range) Normal range of the concentration of the BUN is 2.86-7.14mmol/L(reference value range)
Adverse Event and Serious Adverse Event | visit1(baseline),visit2(2ed week),visit3(6th week),visit4(12th week)
  Safety index

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Feng Liu, MD, Principal Investigator — Second Affiliated Hospital of Soochow University

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make individual participant data (IPD) available to the other researchers, who participant in the study, since this is a muti-center study. The study protocol, statistical Analysis Plan (SAP), informed Consent Form (ICF), clinical Study Report (CSR) will be shared. And all the data collected by the single center will be reported back.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The additional supporting information is shared during the whole period. The IPD will become available immediately after publication.
Access Criteria: Access of the IPD and any additional supporting information will be approved by the principal investigator

REFERENCES:
- [Background] Fasano A, Daniele A, Albanese A. Treatment of motor and non-motor features of Parkinson's disease with deep brain stimulation. Lancet Neurol. 2012 May;11(5):429-42. doi: 10.1016/S1474-4422(12)70049-2. PMID 22516078
- [Background] Reijnders JS, Ehrt U, Weber WE, Aarsland D, Leentjens AF. A systematic review of prevalence studies of depression in Parkinson's disease. Mov Disord. 2008 Jan 30;23(2):183-9; quiz 313. doi: 10.1002/mds.21803. PMID 17987654
- [Background] Chaudhuri KR, Healy DG, Schapira AH; National Institute for Clinical Excellence. Non-motor symptoms of Parkinson's disease: diagnosis and management. Lancet Neurol. 2006 Mar;5(3):235-45. doi: 10.1016/S1474-4422(06)70373-8. PMID 16488379
- [Background] Chaudhuri KR, Schapira AH. Non-motor symptoms of Parkinson's disease: dopaminergic pathophysiology and treatment. Lancet Neurol. 2009 May;8(5):464-74. doi: 10.1016/S1474-4422(09)70068-7. PMID 19375664
- [Background] Yong MH, Fook-Chong S, Pavanni R, Lim LL, Tan EK. Case control polysomnographic studies of sleep disorders in Parkinson's disease. PLoS One. 2011;6(7):e22511. doi: 10.1371/journal.pone.0022511. Epub 2011 Jul 22. PMID 21799880
- [Background] Zesiewicz TA, Sullivan KL, Arnulf I, Chaudhuri KR, Morgan JC, Gronseth GS, Miyasaki J, Iverson DJ, Weiner WJ; Quality Standards Subcommittee of the American Academy of Neurology. Practice Parameter: treatment of nonmotor symptoms of Parkinson disease [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2010 Mar 16;74(11):924-31. doi: 10.1212/WNL.0b013e3181d55f24. PMID 20231670
- [Background] Ashton AK, Jamerson BD, L Weinstein W, Wagoner C. Antidepressant-related adverse effects impacting treatment compliance: Results of a patient survey. Curr Ther Res Clin Exp. 2005 Mar;66(2):96-106. doi: 10.1016/j.curtheres.2005.04.006. PMID 24672116
- [Background] Lam RW. Addressing circadian rhythm disturbances in depressed patients. J Psychopharmacol. 2008 Sep;22(7 Suppl):13-8. doi: 10.1177/0269881108092591. PMID 18753278
- [Background] Hogl B, Arnulf I, Comella C, Ferreira J, Iranzo A, Tilley B, Trenkwalder C, Poewe W, Rascol O, Sampaio C, Stebbins GT, Schrag A, Goetz CG. Scales to assess sleep impairment in Parkinson's disease: critique and recommendations. Mov Disord. 2010 Dec 15;25(16):2704-16. doi: 10.1002/mds.23190. PMID 20931631
- [Background] Ensrud KE, Joffe H, Guthrie KA, Larson JC, Reed SD, Newton KM, Sternfeld B, Lacroix AZ, Landis CA, Woods NF, Freeman EW. Effect of escitalopram on insomnia symptoms and subjective sleep quality in healthy perimenopausal and postmenopausal women with hot flashes: a randomized controlled trial. Menopause. 2012 Aug;19(8):848-55. doi: 10.1097/gme.0b013e3182476099. PMID 22433978
- [Background] Schrag A, Barone P, Brown RG, Leentjens AF, McDonald WM, Starkstein S, Weintraub D, Poewe W, Rascol O, Sampaio C, Stebbins GT, Goetz CG. Depression rating scales in Parkinson's disease: critique and recommendations. Mov Disord. 2007 Jun 15;22(8):1077-92. doi: 10.1002/mds.21333. PMID 17394234
- [Background] Leentjens AF, Verhey FR, Luijckx GJ, Troost J. The validity of the Beck Depression Inventory as a screening and diagnostic instrument for depression in patients with Parkinson's disease. Mov Disord. 2000 Nov;15(6):1221-4. doi: 10.1002/1531-8257(200011)15:63.0.co;2-h. PMID 11104209
- [Background] Richard IH, McDermott MP, Kurlan R, Lyness JM, Como PG, Pearson N, Factor SA, Juncos J, Serrano Ramos C, Brodsky M, Manning C, Marsh L, Shulman L, Fernandez HH, Black KJ, Panisset M, Christine CW, Jiang W, Singer C, Horn S, Pfeiffer R, Rottenberg D, Slevin J, Elmer L, Press D, Hyson HC, McDonald W; SAD-PD Study Group. A randomized, double-blind, placebo-controlled trial of antidepressants in Parkinson disease. Neurology. 2012 Apr 17;78(16):1229-36. doi: 10.1212/WNL.0b013e3182516244. Epub 2012 Apr 11. PMID 22496199
- [Background] Barone P, Poewe W, Albrecht S, Debieuvre C, Massey D, Rascol O, Tolosa E, Weintraub D. Pramipexole for the treatment of depressive symptoms in patients with Parkinson's disease: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2010 Jun;9(6):573-80. doi: 10.1016/S1474-4422(10)70106-X. Epub 2010 May 7. PMID 20452823
- [Result] San L, Arranz B. Agomelatine: a novel mechanism of antidepressant action involving the melatonergic and the serotonergic system. Eur Psychiatry. 2008 Sep;23(6):396-402. doi: 10.1016/j.eurpsy.2008.04.002. Epub 2008 Jun 25. PMID 18583104
- [Result] Rivara S, Mor M, Bedini A, Spadoni G, Tarzia G. Melatonin receptor agonists: SAR and applications to the treatment of sleep-wake disorders. Curr Top Med Chem. 2008;8(11):954-68. doi: 10.2174/156802608784936719. PMID 18673165
- [Result] Lemoine P, Guilleminault C, Alvarez E. Improvement in subjective sleep in major depressive disorder with a novel antidepressant, agomelatine: randomized, double-blind comparison with venlafaxine. J Clin Psychiatry. 2007 Nov;68(11):1723-32. doi: 10.4088/jcp.v68n1112. PMID 18052566